CLINICAL TRIAL: NCT03991091
Title: Reducing Neonatal Morbidity by Discontinuing Oxytocin During the Active Phase of 1st Stage of Labor: a Multicenter Randomized Controlled Trial
Brief Title: Reducing Neonatal Morbidity by Discontinuing Oxytocin During the Active Phase of 1st Stage of Labor
Acronym: STOPOXY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP180581
Record Dates: First submitted 2019-05-24; First posted 2019-06-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Neonatal Morbidity
Keywords: Multicenter; randomized; control study; Oxytocin discontinuation; Neonatal acidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- discontinuation of oxytocin administration (Experimental): Discontinuation of oxytocin administration at the beginning of the active phase of the 1st stage of labor, i.e. oxytocin infusion will be stopped beyond a cervical dilatation of 6cm
  Interventions: Drug: discontinuation of oxytocin administration
- continuation of oxytocin administration (Active Comparator): Standard care in France, i.e. when oxytocin is started during the latent phase of the 1st stage, administration of oxytocin is continued during the active 1st stage and during the 2nd stage if the fetal heart rate is reassuring.
  Interventions: Drug: continuation of oxytocin administration

INTERVENTIONS:
Drug: discontinuation of oxytocin administration — Discontinuation of oxytocin administration at the beginning of the active phase of the 1st stage of labor, i.e. oxytocin infusion will be stopped beyond a cervical dilatation of 6cm. In the experimental group, oxytocin can be re-started, if necessary, after 2 hours of arrest of labor.
  Arms: discontinuation of oxytocin administration
Drug: continuation of oxytocin administration — continuation of oxytocin administration
  Arms: continuation of oxytocin administration

SUMMARY:
The purpose of this study is to measure the impact of a discontinuous administration of oxytocin during the active phase of the 1st stage of labor on the neonatal morbidity rate.

The investigators hypothesize that discontinuation of oxytocin in the active phase of labor (from 6 cm) in women who received oxytocin in the latent phase or for an induction (before 4 cm of dilation) could reduce neonatal morbidity.

DETAILED DESCRIPTION:
Oxytocin is effective in increasing frequency and intensity of uterine contractions and therefore in reducing the duration of labor. Nevertheless, its administration is potentially associated with fetal and maternal short-and long- term complications, such as neonatal acidosis and post-partum hemorrhage and its effectiveness in decreasing caesarean section rate has not been clearly demonstrated.

The most important side effect of oxytocin infusion is uterine hyper-stimulation, which has been shown to occur in more than 30% of women induced with oxytocin. By causing uterine hyper-stimulation, oxytocin infusion may lead to or aggravate abnormal fetal heart rate, contributing to neonatal acidosis. Acidosis is a major part of neonatal morbidity due to related complications such as hospitalization in neonatal intensive care units, but also neonatal death or cerebral palsy in the most severe cases.

The first stage of labor is divided into two phases, a latent phase where cervical dilation is relatively slow until 5-6 cm and an active phase until full dilatation, where cervical dilation accelerates. Currently in France, when oxytocin administration has been initiated during the latent phase, the standard care is to continue it during the whole duration of labor. One assumption is that, once women requiring oxytocin during the latent phase enter the active phase, natural oxytocin takes over from synthetic oxytocin. Thus, in the active phase, oxytocin could be discontinued, reducing exposure duration and therefore reducing the risk of complications, in particular neonatal complications, without compromising the chances of vaginal delivery.

It can therefore be hypothesized that discontinuation of oxytocin in the active phase of labor (from 6 cm) in women who received oxytocin in the latent phase or for an induction (before 4 cm of dilation) could reduce neonatal morbidity.

Several small trials attempting to evaluate this practice have been published, but their design and small population did not allow evaluating the impact of discontinuation of oxytocin on neonatal morbidity. Thus, the investigators propose to conduct a large randomized controlled trial, STOPOXY, aiming to reduce oxytocin exposure and its adverse effects.

The investigators expect an improvement of child health at birth, with less severe neonatal morbidity that may cause neurologic damages and less moderate neonatal morbidity that may be associated with the need of resuscitation and hospitalization.

The investigators plan to conduct a multicenter, randomized, open-label, controlled trial comparing neonatal and maternal outcomes among term singleton neonates after discontinuation or continuation of oxytocin infusion during the active phase of the 1st stage of labor.

Two arms:

* Experimental group: discontinuation of oxytocin administration at the beginning of the active phase of the 1st stage of labor, i.e. oxytocin infusion will be stopped beyond a cervical dilatation of 6cm. In the experimental group, oxytocin can be re-started, if necessary, after 2 hours of arrest of labor.
* Control group: standard care in France, i.e. when oxytocin is started during the latent phase of the 1st stage, administration of oxytocin is continued during the active 1st stage and during the 2nd stage if the fetal heart rate is reassuring.

The open-label design was chosen for several reasons. The main reason is that in case of a blinded trial, the need for un-blinding would be too frequent as the investigators estimate it from the previous published trials at 30 to 40%. The second reason is feasibility. Indeed, in case of non-reassuring fetal heart rate, it is important for the obstetrician to be able to stop the oxytocin infusion to reduce the uterine contractility.

ELIGIBILITY:
Inclusion Criteria:

* With a term (≥37 WG) pregnancy
* Singleton pregnancy
* Fetus in cephalic presentation
* Women receiving oxytocin during the latent phase of the 1st stage of labor, before 4 cm of cervical dilatation, including women with an induction of labor using cervical ripening or oxytocin
* Speaking and reading French language
* Affiliated to social security
* Who have signed the consent form

Exclusion Criteria:

* Women with a scarred uterus
* Fetus with a congenital anomaly
* Fetal growth retardation <3rd percentile
* Having an abnormal fetal heart rate at randomization
* Maternal age < 18 years
* Participating in another trial involving medication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2459 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
neonatal morbidity composite measure | At birth
  Neonatal morbidity will be assessed using a composite variable defined by: an umbilical arterial pH at birth <7.10 and/or a base excess >10mmol/L and/or umbilical arterial lactates>7 mmol/L and/or a 5 minutes Apgar score <7 and/or admission in neonatal intensive care unit (NICU). This composite outcome is based on pertinent and previously published thresholds to assess neonatal acidosis[16]

SECONDARY OUTCOMES:
umbilical cord pH<7.20 | At birth
  umbilical arterial cord pH at birth less than 7.20
umbilical cord pH<7.10 | At birth
  umbilical arterial cord pH at birth less than 7.10
umbilical cord pH<7.00 | At birth
  umbilical arterial cord pH at birth less than 7.00
Need for hypothermia | At birth
  need for hypothermia
other neonatal complications: | 2 hours postpartum
  need of resuscitation at birth
neonatal admission | 2 hours postpartum
  transfer to neonatal care unit
length of the newborn's hospital stay | 0-1 month
  length of hospital stay
mode of delivery | 0-48hours
  cesarean rate
mode of delivery | 0-48hours
  cesarean rate for abnormal fetal heart rate
mode of delivery | 0-48hours
  instrumental vaginal delivery
mode of delivery | 0-48hours
  instrumental delivery for abnormal fetal heart rate
labor duration | 0-48hours
  labor duration (active 1st stage, passive and active 2nd stage)
uterine hyper-stimulation | 0-48hours
  uterine hyper-stimulation, defined by periods with more than 5 uterine contractions in 10 minutes during labor
fetal scalp blood testing | 0-48hours
  need for fetal scalp blood testing during labor
fetal occipito-posterior position | 0-48hours
  fetal occipito-posterior position
maternal hyperthermia | 0-48hours
  maternal fever during labor, defined by maternal temperature >38°C
postpartum hemorrhage | 0-48hours
  post-partum hemorrhage, defined by an estimated blood loss >500mL
The post-partum women's satisfaction | 0 5 day
  women's satisfaction is recorded using the "labor agentry scale". Scores on the Labor Agentry Scale range from 29 to 203, with higher scores indicating greater perceived control during childbirth.
The post-partum women's satisfaction: labor agentry scale | at 2 months postpartum in a survey
  women's satisfaction is recorded using the "labor agentry scale"[18]
The post-partum women's satisfaction | at 2 months postpartum in a survey
  Edinburgh Postnatal Depression Scale. Scores on the Edinburgh Postnatal Depression Scale rabge from 0 to 30, with higher score indicating mental health issues.
The post-partum women's satisfaction | at 2 months postpartum in a survey
  Satisfactiuon of labor and childbirth with Labor Agentry Scale
The post-partum women's satisfaction | at 2 months postpartum in a survey
  Birth experience and well being with EPDS at 2 months
The post-partum women's satisfaction | at 2 months postpartum in a survey
  Breastfeeding at 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Camille Le Ray, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- hospital Cochin; port royal Maternity unit, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Girault A, Sentilhes L, Desbriere R, Berveiller P, Korb D, Bertholdt C, Carrara J, Winer N, Verspyck E, Boudier E, Barjat T, Levy G, Roth GE, Kayem G, Massoud M, Bohec C, Guerby P, Azria E, Blanc J, Heckenroth H, Rousseau J, Garabedian C, Le Ray C; collaborators of the STOPOXY trial and the Groupe de Recherche en Obstetrique et Gynecologie (GROG). Impact of discontinuing oxytocin in active labour on neonatal morbidity: an open-label, multicentre, randomised trial. Lancet. 2023 Dec 2;402(10417):2091-2100. doi: 10.1016/S0140-6736(23)01803-2. Epub 2023 Nov 9. PMID 37952548
- [Result] Girault A, Goffinet F, Le Ray C; collaborators of the STOPOXY trial and the Groupe de Recherche en Obstetrique et Gynecologie (GROG). Reducing neonatal morbidity by discontinuing oxytocin during the active phase of first stage of labor: a multicenter randomized controlled trial STOPOXY. BMC Pregnancy Childbirth. 2020 Oct 20;20(1):640. doi: 10.1186/s12884-020-03331-x. PMID 33081758